CLINICAL TRIAL: NCT06799949
Title: The Role of Endogenous Heparinization As an Intraoperative Predictive Marker for Postoperative ICU Admission: a Prospective Observational Study
Brief Title: The Role of Endogenous Heparinization As an Intraoperative Predictive Marker for Postoperative ICU Admission
Status: Active, not recruiting | Type: Observational
Sponsor: Kotoulas Serafeim-Chrysovalantis (Other)
Responsible Party: Sponsor-Investigator, Kotoulas Serafeim-Chrysovalantis, Principal Investigator, Ippokrateio General Hospital of Thessaloniki
Organization: Ippokrateio General Hospital of Thessaloniki (Other)
Other Study IDs: Ε.Σ.: 842 / 14-01-2025
Record Dates: First submitted 2025-01-24; First posted 2025-01-29 (Actual); Last update posted 2025-02-07 (Actual); Status verified 2025-01

CONDITIONS: Heparinization
Keywords: Endogenous Heparinization; Predictive Marker; Postoperative ICU Admission; Prospective Observational Study; Endothelial Glycocalyx; ROTEM; Major Surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Biospecimen Retention: Samples Without DNA — Blood samples for ROTEM (TEM Innovations GmbH, Munich, Germany) assays
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Adult patients undergoing elective or urgent major abdominal surgeries: * Inclusion Criteria:
    1. Adult patients (>18 years old) undergoing elective or urgent major abdominal surgeries.
    2. ASA ≥ II and/or Surgical Risk score ≥ III
    3. The attending anesthetist's opinion
  * Exclusion Criteria:
    1. Emergency surgeries where preoperative anticoagulant/antiplatelet discontinuation guidelines were not followed.
    2. Patients with liver cirrhosis, trauma and sepsis.
    3. Pregnant or women on reproductive age.
    4. Children
    5. Neurosurgical, cardiovascular and transplantation procedures
    6. Patient's refusal to participate
  Interventions: Diagnostic Test: ROTEM (TEM Innovations GmbH, Munich, Germany) assay

INTERVENTIONS:
Diagnostic Test: ROTEM (TEM Innovations GmbH, Munich, Germany) assay — For each patient, two samples will be collected for ROTEM analysis: one at the beginning of the surgery, during the placement of the arterial line (Start ratio), and another one, at the end, during the completion of the surgical wound closure (Final ratio). The arterial line system will be filled with normal saline (0.9% sodium chloride) without the addition of unfractionated heparin. To avoid sample contamination before sampling, a volume of blood equivalent to 5.5-6 times the dead space (calculated from the catheter tip to the three-way stopcock device) will be aspirated. Blood samples for testing will be stored in specific empty coagulation test tubes (Jiangsu Rongye Technology Co., Ltd, Jiangsu, China) and gently mixed with 3.2%-0.109M sodium citrate, for a total volume of 1.8 ml.

SUMMARY:
This prospective observational study investigates the role of endogenous heparinization as a predictive indicator for postoperative ICU admission. The phenomenon of endogenous heparinization is well documented with growing literature, investigating its clinical significance. The mechanisms leading to the pathogenesis of endogenous heparinization are the following: 1) Liver insufficiency in clearing circulating glycosaminoglycans (GAGs) due to acute liver failure, 2) Neutrophil-induced damage to hepatocytes, which results in releasing sulfated heparan, 3) Direct release of GAGs due to degradation of the endothelial glycocalyx. Furthermore, the endothelial glycocalyx shedding in response to pathological insults such as sepsis, ischemia-reperfusion injury, hyperglycemia, or trauma leads to increased vascular permeability, impaired microcirculation and systemic inflammation. This degradation is associated with several critical conditions, including acute kidney injury, cardiovascular diseases, and multi-organ failure, making glycocalyx shedding a crucial biomarker and therapeutic target. The aim of the study is to evaluate the correlation between intraoperative heparinization through the INTEM/HEPTEM ratio, as an indirect marker of endothelial glycocalyx integrity, and consequently, a biomarker of the patients' physiological status.

DETAILED DESCRIPTION:
This prospective study will include all adult patients scheduled for an elective or urgent major abdominal surgery, who are going to be evaluated preoperatively in our center (Ippokrateio General Hospital of Thessaloniki) The study will be conducted in compliance with ethical standards (Declaration of Helsinki) and has already obtained the approval of the scientific council (Ethics Committee) of our hospital. For every patient informed consent will be obtained. The justification of the request for preoperative ICU bed reservation is going to be based on three criteria: patient's ASA classification, the Surgical Risk score and the attending anaesthetist's opinion and clinical judgment. Patients undergoing neurosurgical, cardiovascular and transplantation procedures will be excluded. All patients will follow the preoperative anticoagulation/antiplatelet discontinuation guidelines. Patients' demographic data, medical history and the necessary laboratory evaluation will be recorded. On the day of the operation the standard anesthetic protocol according to the type of the surgery will be followed and the ESAIC (European Society of Anaesthesia and Intesive Care) standard monitoring will be deployed. All patients are going to receive general anaesthesia. The use of locoregional anaesthesia (epidural, spinal, combined and nerve blocks) mechanical ventilation parameters, hemodynamic parameters, fluid management, ABG analysis results will be recorded in a thorough manner. After anaesthesia induction an arterial line will be placed for direct measurement of arterial pressure, blood gas monitoring of the patient, and simultaneous collection of samples for ROTEM (TEM Innovations GmbH, Munich, Germany) assays. For each patient, two samples will be collected for ROTEM analysis: one at the beginning of the surgery during the placement of the arterial line (Start ratio) and another at the end during the completion of the surgical wound closure(Final ratio). The arterial line system will be filled with normal saline (0.9% sodium chloride) without the addition of unfractionated heparin. To avoid sample contamination before sampling, a volume of blood equivalent to 5.5-6 times the dead space (calculated from the catheter tip to the three-way stopcock device) will be aspirated. Blood samples for testing will be stored in specialized evacuated coagulation test tubes (Jiangsu Rongye Technology Co., Ltd, Jiangsu, China) and gently mixed with 3.2%-0.109M sodium citrate, for a total volume of 1.8 ml. At the end of the surgery, the decision for the patient's postoperative ICU admission will be based on those criteria

* Mental status: Awake and cooperative.
* Oxygenation: PaO₂/FiO₂ ratio ≥ 150-200.
* Ventilation: PaCO₂ < 50 mmHg or baseline.
* RSBI<105.
* Respiratory effort: Spontaneous breathing, no excessive work of breathing.
* Cardiovascular:HR < 140/min; SBP 90-160 mmHg with minimal to no vasopressors.
* Neuromuscular function: TOF ratio ≥ 0.9.
* Attending anaesthetist's opinion and clinical judgement In case of the patients' successful extubation, the risk of re-intubation will be monitored for 24 hours.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (>18 years old) undergoing elective or urgent major abdominal surgery.
* ASA ≥ II and/or Surgical Risk score ≥ III
* The attending anesthetist's opinion

Exclusion Criteria:

* Emergency surgeries where preoperative anticoagulant/antiplatelet discontinuation guidelines were not followed.
* Patients with liver cirrhosis, trauma and sepsis.
* Pregnant or women on reproductive age.
* Children
* Neurosurgical, cardiovascular and transplantation procedures
* Patient's refusal to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 50 patients who will fulfill all the above mentioned inclusion criteria and none of the above mentioned exclusion criteria, will be included in the study. Furthermore, when a patient will meet those criteria a random number generator which will produce only two results (0/1) will be used to decide whether a patient will be included in the study or not.
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2025-01-14 (Actual); Primary Completion 2025-04-30 (Estimated); Study Completion 2025-04-30 (Estimated)

PRIMARY OUTCOMES:
Need for Postoperative ICU Admission | 24 hours
  At the end of the surgery, the decision for the patient's postoperative ICU admission will be based on commonly used criteria in clinical practice and the Anesthesiology, who will decide that will be blinded to the research.

CONTACTS AND LOCATIONS:
Locations (1):
- Ippokrateio General Hospital of Thessaloniki, Thessaloniki, Thessaloniki, Greece

IPD SHARING:
Plan to Share IPD: Yes
Raw data with no individual-identifying information
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: The IPD and supporting information will be available after the publication of the results of the study, which is expected to take place within 2025, with no expiration date.
Access Criteria: The IPD and supporting information will be accessible to everyone, upon request to the leading author of the publication that will result from this study